CLINICAL TRIAL: NCT04968548
Title: Determination and Validation of Lung EpiCheck®: A Multianalyte Assay for Lung Cancer Prediction. A Case-Control Study
Brief Title: Determination and Validation of a Multi-analyte Assay for Lung Cancer Screening
Status: Active, not recruiting | Type: Observational
Sponsor: Nucleix Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Lung-RND-003
Record Dates: First submitted 2021-07-04; First posted 2021-07-20 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Lung Cancer
Keywords: LDCT; Low Dose CT; Lung Cancer Screening; liquid biopsy; early detection; lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases Series: Subjects with confirmed lung cancer diagnosis
  Interventions: Procedure: Blood collection
- Screening Series: Subjects undergoing LDCT for lung cancer screening
  Interventions: Procedure: Blood collection

INTERVENTIONS:
Procedure: Blood collection — Peripheral blood will be collected via routine venipuncture procedure

SUMMARY:
This study is part of the development and validation of a non-invasive lung screening test which aim to identify early stage lung cancer in patients at high risk for lung cancer.

DETAILED DESCRIPTION:
This is a prospective, case-control, multi-center, observational nonsignificant risk study. The study aims to collect blood and clinical data from subjects undergoing Low Dose CT (LDCT) for lung cancer screening and subjects with confirmed lung cancer.

ELIGIBILITY:
Inclusion Criteria - Cases:

* Current or past smokers, with at least 20 pack-years
* Subjects with either A high suspicion for lung cancer, with planned surgery to establish a definitive diagnosis within 60 days after date of blood collection OR treatment naive lung cancer patients

Exclusion Criteria - Cases:

* Known diagnosis or treatment of any previous cancer, including lung cancer, in the past 5 years, except for fully resected non-melanoma skin cancer or fully-resected carcinoma in situ of the cervix
* Current lung cancer is known to be stage III or IV by pathology.

Inclusion Criteria - Screening:

- Current or past smokers, with at least 20 pack-years, undergoing LDCT for lung cancer screening

Exclusion Criteria - Screening:

* Known diagnosis or treatment of any cancer, including lung cancer, in the past 5 years, except for fully resected non-melanoma skin cancer or fully-resected carcinoma in situ of the cervix
* Subjects whose purpose of performing LDCT is for surveillance of a lung nodule

Ages: 50 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The Case Series will include subjects 50-80 years old, current or past smokers with at least 20 pack-years, with either (a) a high suspicion for lung cancer, who are planning to undergo surgery to establish a definitive diagnosis; or (b) confirmed lung cancer diagnosis, however did not yet undergo any treatment for this cancerous lesion.
  The Screening Series will include subjects 50-80 years old, current or past smokers, with at least 20 pack-years, undergoing LDCT for lung cancer screening.
  All subjects should be without other cancer in the past 5 years except for fully resected non-melanoma skin cancer or fully-resected carcinoma in situ of the cervix
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Collection of blood samples | 24 Months
  Collect blood to support the development and validation of a multi analyte test for lung cancer screening
Clinical data collection | 24 Months
  Collect clinical data to support the development and validation of a multi analyte test for lung cancer screening

SECONDARY OUTCOMES:
Performance | 36 Months
  Performance of the assay in terms of (1) Sensitivity (2) Specificity (3) NPV (negative predictive value) and (4) PPV (positive predictive value)
Sensitivity | 36 Months
  Performance of the assay in terms of Sensitivity
Specificity | 36 Months
  Performance of the assay in terms of Specificity
Negative Predictive Value | 36 Months
  Performance of the assay in terms of NPV (negative predictive value)
Positive Predictive Value | 36 Months
  Performance of the assay in terms of PPV (positive predictive value)

CONTACTS AND LOCATIONS:
Overall Officials: Radha Duttagupta, PhD, Study Director — Nucleix Ltd.
Locations (31):
- United States (27):
  - Scripps Memorial Hospital, Encinitas, California
  - Centura Health, Lakewood, Colorado
  - VA Connecticut Healthcare System, West Haven, Connecticut
  - Orlando Health, Inc., Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - St. Elizabeth Edgewood Hospital, Edgewood, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Owensboro Health, Owensboro, Kentucky
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - University of Minnesota Health, Minneapolis, Minnesota
  - Harry S. Truman Memorial Veterans' Hospital, Columbia, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - Northwell Health, New Hyde Park, New York
  - University of Rochester, Rochester, New York
  - The University of North Carolina, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Durham VA Health Care System, Durham, North Carolina
  - W.G. (Bill) Hefner VA Medical Center, Salisbury, North Carolina
  - Novant Health Cancer Research, Winston-Salem, North Carolina
  - Summa Health, Akron, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Baptist Cancer Center, Memphis, Tennessee
  - Michael E. DeBakey VA Medical Center, Houston, Texas
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - Vancouver General Hospital/The University of British Columbia, Vancouver, British Columbia
  - University Health Network, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaga M, Chorostowska-Wynimko J, Horvath I, Tammemagi MC, Shitrit D, Eisenberg VH, Liang H, Stav D, Levy Faber D, Jansen M, Raviv Y, Panagoulias V, Rudzinski P, Izbicki G, Ronen O, Goldhaber A, Moalem R, Arber N, Haas I, Zhou Q. Validation of Lung EpiCheck, a novel methylation-based blood assay, for the detection of lung cancer in European and Chinese high-risk individuals. Eur Respir J. 2021 Jan 14;57(1):2002682. doi: 10.1183/13993003.02682-2020. Print 2021 Jan. PMID 33122336